CLINICAL TRIAL: NCT07243834
Title: Assessing a Digital Exercise Intervention for Health Outcomes and Engagement in Regular Exercise (ADHERE): A Randomised Controlled Trial Comparing the Efficacy of a Digital Exercise Intervention With Virtual Supervised Group Exercise Sessions to Standard of Care on Exercise Adherence at Six Months in Patients With Prostate Cancer Undergoing Hormone Therapy.
Brief Title: Assessing a Digital Exercise Intervention for Health Outcomes and Engagement in Regular Exercise
Acronym: ADHERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCR6225
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Cancer (Diagnosis)
Keywords: Exercise intervention; physical activity; adherence
MeSH Terms: conditions — Prostatic Neoplasms; Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SoC) (No Intervention): Participants will be sent a link to a webpage which provides information on physical activity and exercise guidelines, local and nationally available exercise, and contact details for the RMH physiotherapy department with the option to self-refer for further support.
- SoC + digital exercise intervention with virtual supervised group exercise sessions (Experimental): Participants will receive standard of care and a digital exercise intervention.
  Interventions: Other: Participation in a digital exercise intervention with virtual supervised group exercise sessions

INTERVENTIONS:
Other: Participation in a digital exercise intervention with virtual supervised group exercise sessions — The intervention will involve an initial individual review with a clinical exercise physiologist (CEP) to complete a screening questionnaire, set goals and discuss details of physical activity and the exercise plan.
  Participants will then attend weekly virtual supervised group exercise sessions and have access to pre-recorded exercise videos as well. Participants will receive motivational emails after each group session and have check-in phone calls with the CEP at week 4 and week 8.
  Participants will also have the option to take part in the patient buddy scheme which includes three support phone calls from a fellow patient at The Royal Marsden NHS Foundation Trust. One phone call will be scheduled at the start of the exercise programme, one halfway through the programme, and one at the end of the programme.
  Individual review appointments with the CEP will be scheduled at Week 13 and Week 26 to review progress and address any barriers to exercise adherence.
  Other Names: Exercise intervention
  Arms: SoC + digital exercise intervention with virtual supervised group exercise sessions

SUMMARY:
Patients diagnosed with prostate cancer and receiving hormone therapy in conjunction with radiotherapy are likely to suffer from adverse effects caused by ADT treatment either short term or long term. The most common side effects include changes in body composition leading to increased visceral fat and reduced lean muscle mass, increased risk of cardiovascular events and fatigue, which overall lower quality of life.

There is strong evidence to support exercise interventions in minimising, and in some cases reversing many ADT -related toxicities, but exercise adherence remains a challenge for people living with prostate cancer, particularly due to logistical barriers to attendance such as cost and travel time, as well as insufficient motivation.

The aim of this single centre, phase III randomised controlled trial is to assess the efficacy of a new digital exercise programme with virtual supervised group exercise sessions in improving adherence to exercise guidelines.

The trial aims to recruit 160 participants with prostate cancer undergoing ADT, who will be allocated either the standard of care group or standard of care plus participation in the digital exercise intervention on a 1:1 ratio.

Adherence to physical activity will be measured using a wearable accelerometer, an exercise diary, self-reported questionnaires and clinic based assessments at 3 months, 6 months and 12 months post radiotherapy treatment. Recruitment will take place at the Royal Marsden NHS Foundation Trust, Chelsea.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 at randomisation
2. Men with histological confirmation of prostate adenocarcinoma who are receiving or planned to receive ADT with an LHRHa as part of their PCa treatment
3. If already started ADT, have received no more than eight weeks ADT at randomisation
4. Planned for radiotherapy
5. Assessed by clinical team to be safe to exercise and safe to enter the trial with no absolute contraindications to exercise as defined by clinical guidance
6. Able to use technological aspects of the intervention including access to MyMarsden and a device for video conferencing
7. Fluent in English and able to understand instructions
8. WHO performance status 0-2
9. Able to give written informed consent

Exclusion Criteria:

1. Men planned to receive an androgen receptor-targeted agent (ARTA) or chemotherapy
2. Absolute contraindication to exercise as defined by ACPICR standards. This includes:

   * New symptoms of angina
   * New or unstable heart failure
   * Newly diagnosed diabetes that is not controlled
   * New or untreated arrhythmias
   * Resting tachycardia or new bradycardia (not linked to changes in medications)
   * Symptomatic hypotension
   * Uncontrolled hypertension (SBP ≥ 180mmHg or DBP≥ 100mmHg)
3. Unstable spinal bone metastasis or at high risk of a fracture
4. Musculoskeletal issue inhibiting exercise

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2030-04-28 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is adherence to physical activity and exercise guidelines assessed using device-based activity data and self-reported physical activity and exercise data at six-months post-radiotherapy. | Measured at six months post radiotherapy
  Activity data will be measured using the ActiGraph LEAP wearable activity monitor and an Exercise Diary.
  To calculate physical activity and exercise adherence, we will compare the measured total volume of physical activity compared to the target volume of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden Hospital, London, United Kingdom